CLINICAL TRIAL: NCT05965830
Title: PRospective Observational Study Comparing Electromyography of the Diaphragm With Ultrasound in Neonates and Children With REspiratory Support: the PROCEDURES Study
Brief Title: Comparing Electromyography of the Diaphragm With Ultrasound in Neonates and Children With Respiratory Support
Acronym: PROCEDURES
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, sgjheisterkamp, Pediatric intensivist, Leiden University Medical Center
Other Study IDs: P23-007
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ultrasound; Transcutaneous EMG; Diaphragm; Neonate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: The study population consists of clinically stable infants or pediatric patients up to 12 months of age admitted to the PICU.
  Interventions: Device: Diaphragm ultrasound

INTERVENTIONS:
Device: Diaphragm ultrasound — A single, simultaneous assessment of the diaphragm muscle functioning through dEMG and dUS at the time of spontaneous breathing.
  Other Names: transcutaneous diaphragm EMG

SUMMARY:
Background of the study:

Increased work of breathing, potentially leading to respiratory insufficiency, resulting in the need of (non-) invasive respiratory support is the most common observed problem in the neonatal - and pediatric intensive care unit (NICU/PICU). The diaphragm is the main respiratory muscle. Currently there is not an established technique accessible to observe the (clinical) function of the diaphragm and its role in respiratory insufficiency. New non-invasive modalities are promising, such as transcutaneous diaphragm electromyography (dEMG) and diaphragm ultrasound (dUS).

Objective of the study:

Our objective is to assess the association between transcutaneous diaphragm electromyography (dEMG) and diaphragm ultrasound (dUS) in the PICU population.

Study design:

Single center pilot study

Study population:

The study population consists of children between 0-12 months, admitted to the PICU of the Leiden University Medical Center, with invasive respiratory support.

Primary study parameters/outcome of the study:

Primary endpoint is to evaluate the association between dEMG and dUS measurements in the PICU population.

DETAILED DESCRIPTION:
All clinically stable infants or pediatric patients up to 12 months of age admitted to the PICU with invasive respiratory support comply with the extubation readiness test (ERT) criteria are included after informed consent. After inclusion simultaneous monitoring of the diaphragm muscle function using transcutaneous diaphragm electromyography (dEMG) and diaphragm ultrasound (dUS) will take place while the patient is on spontaneous breathing mode during ERT.

Transcutaneous diaphragm electromyography measurements are performed using three skin electrodes; two electrodes are bilaterally placed at the costo-abdominal margin in the nipple line and one at or above the sternum during a time period of 15 minutes, with a maximum of 30 minutes.

Ultrasound examination is performed using a linear transducer, and micro-convex transducer by trained operators.

The views are achieved with the patient in supine position. Diaphragm excursion (DE), diaphragm thickness (DT) and diaphragm thickening fraction (DTF) are measured, performed at three different breathing cycles within one examination event.

After completion of the measurements analysis will be performed to evaluate the association between dEMG and dUS outcomes in this specific PICU population.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 - 12 months of age at the moment of inclusion and born ≥ 37 weeks gestational age.
* Specific patients cohort PICU:

pediatric patients with invasive respiratory support comply with the extubation readiness test (ERT) criteria

* No spontaneous breathing for the duration of the assessment
* Written parenteral informed consent (IC)
* A patient can only participate once

Exclusion Criteria:

* Unilateral diaphragm paresis diagnosed by ultrasound
* Congenital malformations not compatible with dEMG
* Need of cardiac pacing
* Congenital muscle atrophy disorder
* Clinical instability requiring frequent interventions by the nursing staff that may interfere with the measurements
* The attending physician considers the patient to be too vulnerable to participate in the study

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of clinically stable infants or pediatric patients up to 12 months of age admitted to the PICU.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-25 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Association between dEMG amplitude and dUS diaphragm thickening fraction and dEMG tonic activity and diaphragm thickness | 1 year
  Evaluation of the association between dEMG and dUS measurements in the PICU population with invasive respiratory support. Pearson's correlation coefficient is used to quantify the correlation between dEMG and dUS variables.

SECONDARY OUTCOMES:
Assessment of patient specific values of dEMG and dUS | 1 year
  To assess patient specific values of dEMG and dUS measurements in the PICU population while on spontaneous breathing

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Intensive Care Unit, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided